CLINICAL TRIAL: NCT04510831
Title: Measuring Dietary Iron Absorption From Edible Insects and Assessing the Effect of Chitin Content on Iron Bioavailability: Stable Iron Isotope Studies in Young Women (Study 1, Tenebrio Molitor)
Brief Title: Measuring Dietary Iron Absorption From Edible Insects and Assessing the Effect of Chitin Content on Iron Bioavailability (Study 1)
Acronym: Sustironable1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Zurich University of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: Sust-iron-able1
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Iron-deficiency
Keywords: chitin; iron deficiency; Tenebrio molitor; iron bioavailability; edible insects
MeSH Terms: conditions — Anemia, Iron-Deficiency; Iron Deficiencies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Refined maize (Experimental): Two portions of porridge prepared with refined maize flour with extrinsic addition of labelled FeSO4 (isotopic iron 54)
  Interventions: Other: Refined maize with extrinsic addition of labelled FeSO4
- T.molitor native chitin (Experimental): Two portions of porridge prepared with refined maize flour mixed with dried intrinsically labelled Tenebrio molitor (isotopic iron 57) native chitin and extrinsic addition FeSO4 (isotopic iron 58)
  Interventions: Other: T.molitor native chitin
- T.molitor reduced chitin (Experimental): Two portions of porridge prepared with refined maize flour mixed with dried intrinsically labelled Tenebrio molitor (isotopic iron 57) reduced chitin and extrinsic addition FeSO4 (isotopic iron 58)
  Interventions: Other: T molitor reduced chitin

INTERVENTIONS:
Other: Refined maize with extrinsic addition of labelled FeSO4 — Porridge prepared with refined maize flour with extrinsic addition of FeSO4 (isotopic iron 54)
  Arms: Refined maize
Other: T.molitor native chitin — Porridge prepared with dried intrinsically labelled T.molitor (isotopic iron 57) native chitin, refined maize flour and extrinsic addition FeSO4 (isotopic iron 58)
  Arms: T.molitor native chitin
Other: T molitor reduced chitin — Porridge prepared with dried intrinsically labelled T.molitor (isotopic iron 57) reduced chitin, refined maize flour and extrinsic addition FeSO4 (isotopic iron 58)
  Arms: T.molitor reduced chitin

SUMMARY:
Due to the growing world population, there is a need to develop viable ecological and nutritional alternatives to animal food products. However, animal products are a key dietary source of well-absorbed iron, and iron deficiency and iron deficiency anemia remain highly prevalent in high- and low-income countries. Meat and fish provide a substantial proportion of absorbed iron in the western diet by two distinct components: a) heme iron is well absorbed (20-45% fractional absorption) and is not affected by most dietary enhancers and inhibitors, which often affect non-heme iron absorption; b) peptides in muscle meat exert an enhancing effect the absorption of non-heme iron contained in other meal components. The potential of edible insects as a dietary source of well-absorbed iron has not been investigated in detail. In particular, it is unclear whether insects provide an iron moiety similar to hemoglobin which would be well absorbed and unaffected by other dietary components, and whether their presence in a test meal exerts an enhancing effect on iron bioavailability from the whole meal.

Furthermore, chitin, a major component of insect biomass, is a known iron binder and is potentially responsible for a decreased iron absorption from insect-based foods. Decreasing chitin content could allow the high amounts of iron in insects to be well-absorbed, and enhance the absorption of iron from plant-based foods. To differentiate iron absorption from insect biomass from other sources, insects will be intrinsically labelled with the stable iron isotope 57Fe, while other food iron components will be labelled with the iron isotope 58Fe.The present study will provide novel data to elucidate the nutritional value as sources of dietary iron of insect species (Tenebrio molitor). Since 2017 T.molitor is recognised as an edible insect in the Swiss food legislation and commercially available (Essento Food AG, Zürich; Insekterei, GmbH, Zürich).

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 to 45 years old
* Normal Body Mass Index (18.5 - 25 kg/m2)
* Body weight ≤ 65 kg
* Non-anemic (hemoglobin (Hb) >12.0 g/dL)
* Low iron status (being in the lower half of the serum ferritin distribution at screening)
* Normal CRP (<5.0 mg/L), indicating no inflammation
* Knowledge of English at least at level B2 (assessed by self-declaration)
* Signed informed consent

Exclusion Criteria:

* Pregnancy (assessed by self-declaration)
* Lactating up to 6 weeks before study initiation
* Any metabolic, gastrointestinal kidney or chronic disease such as diabetes, hepatitis, hypertension, cancer or cardiovascular diseases (according to the participants own statement)
* Continuous/long-term use of medication (except for oral contraceptives and anti-acne medication)
* Consumption of mineral and vitamin supplements within 2 weeks prior to 1st meal administration
* Blood transfusion, blood donation or significant blood loss (accident, surgery) over the past 4 months
* Earlier participation in a study using iron stable isotopes or participation in any clinical study within the last 30 days
* Participant who cannot be expected to comply with study protocol e.g. not available on certain study appointments
* Cigarette smoking ( > 1 cigarette per day)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2020-12-09 (Actual)

PRIMARY OUTCOMES:
Fractional Iron absorption | 30th day of the study
  Fractional iron absorption will be calculated based on the shift of the iron isotope ratios in the collected blood samples after the administration of the intervention products .Fractional iron absorption will be measured as erythrocyte incorporation of the naturally occurring iron forms with different masses used to label the iron supplements.

SECONDARY OUTCOMES:
Hemoglobin (Hb) | screening (-1), day 16th and day 30th of the study
  Iron status marker
Plasma ferritin (PF) | screening (-1), day 16th and day 30th of the study
  Iron status marker
C-Reactive Protein (CRP) | screening (-1), day 16th and day 30th of the study
  Inflammation status
Soluble transferring receptor (sTfR) | screening (-1), day 16th and day 30th of the study
  Iron status marker
Body iron stores (BIS) | screening (-1), day 16th and day 30th of the study
  Iron status marker
Alpha 1 acid glycoprotein (AGP) | screening (-1), day 16th and day 30th of the study
  Inflammation marker

CONTACTS AND LOCATIONS:
Overall Officials: Nikolin Hilaj, MSc, Principal Investigator — Laboratory of Human Nutrition ETH Zürich
Locations (1):
- ETH Zurich, Laboratory of Human Nutrition, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hilaj N, Zimmermann MB, Galetti V, Zeder C, Murad Lima R, Hammer L, Krzystek A, Andlauer W, Moretti D. The effect of dechitinization on iron absorption from mealworm larvae (Tenebrio molitor) flour added to maize meals: stable-isotope studies in young females with low iron stores. Am J Clin Nutr. 2022 Oct 6;116(4):1135-1145. doi: 10.1093/ajcn/nqac210. PMID 36100966